CLINICAL TRIAL: NCT03298490
Title: Reliability, Validity Of The Turkish Version Of The Back Performance Scale
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, GÖKHAN MARAŞ, Research assistant, Gazi University
Other Study IDs: 2017-73
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain
Keywords: validity; reliability; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we performed the validity and reliability of the Turkish version of Back Performance Scale.

DETAILED DESCRIPTION:
Low back pain (LBP) is defined as the pain that occurs in the area between the lower border of the scapula and the buttocks and sometimes radiates to the lower extremities. In the community, lower back pain is the second most common health problem after cold. 15% of LBP cases are chronic. Appropriate use of assessment questionnaires is one of the most important steps in the evaluation of the functional level of the patient and in deciding on an effective treatment protocol. The purpose of study is to determine the Turkish version, validity and reliability of Back Performance Scale. 180 patients with chronic low back pain were included in the study. Test-retest and internal consistency analysis were conducted to determine the reliability of the questionnaire. Test-retest results evaluated using the Intraclass Correlation Coefficient method.

ELIGIBILITY:
Inclusion Criteria:

* Having a low back pain
* Literate persons

Exclusion Criteria:

* Cancer disease
* Trauma
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic back pain between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
Roland Morris disability questionnaire | 10 minute
  Roland Morris Disability Questionnaire, a widely used health status measure for low back pain. The RMDQ can be used in research or clinical practice.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 10 minute
  The Oswestry Disability Index (ODI) has become one of the principal condition-specific outcome measures used in the management of spinal disorders

CONTACTS AND LOCATIONS:
Overall Officials: seyit çıtaker, Study Chair — gazi üniversity
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)